CLINICAL TRIAL: NCT03919513
Title: Effect of Combined Inspiratory Muscle Training and Continuous Positive Airway Pressure in Pulmonary Rehabilitation for Chronic Obstructive Pulmonary Disease.
Brief Title: Effect of Combined IMT and CPAP in Pulmonary Rehabilitation for COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-HXNK-011
Record Dates: First submitted 2019-04-04; First posted 2019-04-18 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2019-01

CONDITIONS: Pulmonary Rehabilitation
Keywords: IMT,NPPV,Pulmonary rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- respiratory muscle weakness (Experimental): Patients with respiratory muscle weakness are performing the inspiratory pressure threshold device, combined CPAP and inspiratory pressure threshold device and continue oxygen therapy randomly.
  Interventions: Device: inspiratory pressure threshold device
- normal respiratory muscle (Experimental): Patients with normal respiratory muscle are performing the inspiratory pressure threshold device, combined CPAP and inspiratory pressure threshold device and continue oxygen therapy randomly.
  Interventions: Device: inspiratory pressure threshold device

INTERVENTIONS:
Device: inspiratory pressure threshold device — The threshold loading device is composed of a mouth -piece attached to a small plastic cylinder that contains a spring-loaded poppet value. The valve opens to permit inspiratory flow only once the person has generated adequate negative intrathoracic pressure to condense the spring.
  Other Names: CPAP

SUMMARY:
Inspiratory muscle training(IMT) was one of the widely used pulmonary rehabilitation method in COPD patients.However, when the respiratory muscles are fatigue without sufficient rest, IMT may increase muscle fatigue and aggravate muscle damage. Noninvasive positive pressure ventilation (NPPV) is another important strategy of pulmonary rehabilitation which could overcome airway resistance and reduce respiratory work, improve respiratory muscle fatigue. Therefore, the purpose of this study was to explore the effective of the "IMT - NPPV sequential" rehabilitation method, that is, first inspiratory muscle training, followed by respiratory muscle resting (non-invasive positive pressure ventilation).

DETAILED DESCRIPTION:
Exploring the effects of the new rehabilitation method of "IMT - NPPV sequential", comparing with the single rehabilitation strategy such as inspiratory muscle training and non-invasive positive pressure ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary function test of forced expiratory volume at one second (FEV1)/forced vital capacity(FVC) < 70% after inhalation of bronchial dilation agent. Patients in a clinically stable state.

Exclusion Criteria:

* Patients were excluded if they had other respiratory diseases ,or evidence of pneumothorax or mediastinal emphysema and pacemaker installed.

Patients with acute cardiovascular event and severe cor pulmonale. Patients with poor compliance. An Other causes of diaphragmatic dysfunction

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength(composite outcome measure) | Change from baseline to 8 weeks
  Currently, the maximal inspiratory pressure (PImax) and maximal expiratory pressures(PEmax) are measured by a digital manometer (AZ-8205, AZ Instrument, Taichung City, Taiwan)and combined to evaluate respiratory muscle function.

SECONDARY OUTCOMES:
Diaphragmatic function | Change from baseline to 8 weeks
  Diaphragmatic function can be assessed by diaphragm electromyogram (EMGdi) measured by a high-performance data acquisition device (Powerlab 16/35; ADInstruments, Australia), which reflect the physiological activity of the diaphragm and indicate functional status of the central drive.
Symptom Evaluation(composite outcome measure) | Change from baseline to 8 weeks
  Individuals with chronic respiratory disease often have symptoms such as dyspnea, fatigue, cough, weakness, sleeplessness, and psychological distress. Instruments for assessment of multiple symptoms include COPD Assessment Test (CAT) and Modified Medical British Research Council Scale(mMRC).
Pulmonary function(composite outcome measure) | Change from baseline to 8 weeks
  Pulmonary function is measured using a spirometer(PonyFX 229, Cosmed, Rome, Italy) that is calibrated daily.The FEV1 and percent-of-predicted FEV1, FVC and percent-of-predicted FVC which are presented in one report are used to evaluate Pulmonary Function.
Exercise capacity | Change from baseline to 8 weeks
  Exercise capacity is evaluated using the 6-min walking distance (6MWD) according to American Thoracic Society guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Xin, Doctor, Principal Investigator — Zhujiang Hospital,Southern Medical Unversity
Locations (1):
- Zhujiang Hospital,Southern Medical Universicity, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No